CLINICAL TRIAL: NCT00688168
Title: Identifying the Role of Inflammatory Cytokines in Symptom Production in Multiple Myeloma
Brief Title: Inflammatory Cytokines in Symptom Production in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007-0612
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Phone Call; Treatment Naive; Inflammatory Cytokines; Questionnaire; Survey; Interactive Voice Response; Symptom Production; Pain; IVR; MM
MeSH Terms: conditions — Multiple Myeloma; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue sample by inserting a swab into mouth and rubbing firmly against the inside of cheeck or underneath lower or upper lip for about a minute during a regularly schedule clinic visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptom Assessments: Patients diagnosed with multiple myeloma (MM) complete questionnaires with Neurocognitive Testing and Neurosensory Testing
  Interventions: Behavioral: Questionnaire; Behavioral: Neurocognitive Testing; Behavioral: Neurosensory Testing

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires measuring pain and other symptoms, mood, and quality of life.
  Other Names: Survey
Behavioral: Neurocognitive Testing — A neurocognitive exam (tests to check your memory and thinking abilities, for example) will be performed.
Behavioral: Neurosensory Testing — Neurosensory testing will be performed to find out how sensitive you are to things such as touch, coolness, warmth, pinprick on the finger, and squeezing of the skin on the finger, hand, or arm.

SUMMARY:
The goal of this research study is to learn about the pain and/or other symptoms that patients may experience either while you are being monitored by your doctor before a decision is made to start you on treatment for your MM, or during and after treatment for MM, and how these symptoms may affect therapy. A second goal is to learn how differences in genes may affect the symptom burden from cancer and cancer therapy.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete 5 questionnaires during a regularly scheduled clinic visit. These questionnaires will measure pain and other symptoms, such as your mood and quality of life. You will also be asked to give a tissue sample by inserting a swab into your mouth and rubbing firmly against the inside of your cheek or underneath your lower or upper lip for about a minute at most. Completing the 5 questionnaires and the swab sample collection takes about 30 minutes in total.

This is an investigational study.

Up to 500 patients will take part in the cross-sectional phase of this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Must speak and understand English;
2. Must be diagnosed with MM and meet one of the following criteria: 1) have been treated for MM with steroids only, or have received no more than two cycles of induction chemotherapy for MM and are going to be treated with bortezomib or thalidomide for induction therapy; 2) have received induction therapy and have been approved (or are being approved) medically and financially to receive autologous hematopoietic stem cell transplantation (Auto-HSCT); 3) cross sectional study patients will be either with a current diagnosis of asymptomatic MM not receiving treatment; or at least 12 months from the MM diagnosis, had received induction therapy, with or without received autologous hematopoietic stem cell transplantation (Auto-HSCT) and follow-up treatments. This cohort for a cross sectional survey may include the cases been enrolled, either completed or dropped from the same study. It may also include patients who did not participate on the first phase of the protocol (longitudinal cohort).
3. Patients >= 18 years old.

Exclusion Criteria:

1. Patients who do not understand the intent of the study, so cannot or will not give informed consent
2. Patients who are unable to use the Interactive Voice Response (IVR) system due to physical limitations (e.g., hearing impairment).
3. Induction therapy patients with a neuropathy score of 3 or greater on the NCI's Common Terminology Criteria (CTC version 3.0) either at the beginning of induction chemotherapy or after 1-2 cycles of chemotherapy as a result of previous treatment or from some other comorbid cause. This exclusion criteria does apply to the auto-HSCT patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, 18 years or older, diagnosed with multiple myeloma (MM).
Sampling Method: Non-Probability Sample
Enrollment: 491 (Actual)
Dates: Start 2008-05-09 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Multiple myeloma module of MDASI (MDASI-MM) Questionnaire | Baseline with 12 Month Longitudinal Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org